CLINICAL TRIAL: NCT06256198
Title: Comparison Between PCO2 Gap, Lactate and Procalcitonin as Predictors of Clinical Outcome in ICU Septic Patients
Brief Title: Role of PCO2 Gap as Predictor of Clinical Outcome in ICU Septic Patients
Acronym: PCO2
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed wagih Ezzat deusouky, lecturer of anesthesia, Ain Shams University
Other Study IDs: MS 719/2022
Record Dates: First submitted 2024-01-31; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: survivors
  Interventions: Other: measurement of serum lactate and procalcitonin and PCO2 gap
- Group M: non survivors
  Interventions: Other: measurement of serum lactate and procalcitonin and PCO2 gap

INTERVENTIONS:
Other: measurement of serum lactate and procalcitonin and PCO2 gap — measurement of serum lactate, procalcitonin and PCO2 gap

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection, if not recognized early and managed promptly, it can lead to septic shock, multiple organ failure and death. Sepsis is associated with high mortality, and the early recognition of the signs of tissue hypo perfusion is crucial in its management.

This prospective study was aimed to detect that PCO2 gap can be taken as a reliable prognostic tool in septic patients

DETAILED DESCRIPTION:
In the community setting, sepsis often presents as the clinical deterioration of common and preventable infections. Sepsis also frequently results from infections acquired in health care settings, which are one of the most frequent adverse events during care delivery and affect hundreds of millions of patients worldwide every year The venous-to-arterial carbon dioxide difference (Pv-aCO2) can indicate the adequacy of microvascular blood flow in the early phases of resuscitation in sepsis. Hence, other resuscitation goals, such as PCO2 gap, have been suggested, due to their ability to predict adverse clinical outcomes and simplicity in patients achieving normal oxygen-derived parameters during the early phases of resuscitation in septic shock.

Blood lactate level is also useful in evaluating sepsis. Serum lactate is a good indicator of the presence of hypoxic tissue during septic shock, since its production takes place during Anerobic metabolism.

Procalcitonin (PCT) is the precursor of calcitonin, and higher levels are associated with the development of sepsis. Com¬monly, there is an elevation of PCT levels 4 h after the on¬set of symptoms, peaking between 8 h and 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Adult septic patients ≥ 21 years old

Exclusion Criteria:

* Patients with history of chronic obstructive pulmonary disease and bronchial asthma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in ICU departments with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
prediction of clinical outcome in ICU septic patients | 48 hours
  PCO2 gap mmHg will be measured on admission and after 48 hours